CLINICAL TRIAL: NCT02119052
Title: Effect of Long-acting Somatostatin on Liver in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Effects of Somatostatin on Liver in ADPKD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ADPKD-liver
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-01

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OCTEOTRIDE (Experimental): octeotride 20 mg, intramuscular injection monthly for 3 years
  Interventions: Drug: octeotride
- Placebo (Placebo Comparator): Placebo (saline soluction), intramuscular injection monthly for 3 years
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: octeotride
  Arms: OCTEOTRIDE
Drug: placebo
  Arms: Placebo

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is associated with the development of a variety of extrarenal manifestations of which polycystic liver disease is most common. The investigators aimed to assess the changes over time of liver volume in ADPKD patients and whether it is affected by the treatment with the somatostatin analogue, octreotide.

35 ADPKD patients (14 males) aged 34±8 years were randomly assigned to 36 month treatment with placebo (n=18) or octreotide (n=17). Clinical and liver parameters at magnetic resonance (RM) were evaluated at baseline, study end and after 24 months of drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of autosomal dominant polycystic kidney and liver disease
* glomerular filtration rate greater than 40 ml/min

Exclusion Criteria:

* diabetes mellitus
* proteinuria greater than 1 g/24 hours
* significant glomerular disease
* urinary tract lithiasis and infections
* symptomatic gallstones
* biliary sludge
* cancer
* pregnant women
* lactanting women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-01; Primary Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Effect of somatostatin on liver volume | 3 years

REFERENCES:
- [Derived] Pisani A, Sabbatini M, Imbriaco M, Riccio E, Rubis N, Prinster A, Perna A, Liuzzi R, Spinelli L, Santangelo M, Remuzzi G, Ruggenenti P; ALADIN Study Group. Long-term Effects of Octreotide on Liver Volume in Patients With Polycystic Kidney and Liver Disease. Clin Gastroenterol Hepatol. 2016 Jul;14(7):1022-1030.e4. doi: 10.1016/j.cgh.2015.12.049. Epub 2016 Feb 1. PMID 26844873